CLINICAL TRIAL: NCT02709564
Title: Single Dose Versus Two Doses of Sublingual Misoprostol in Decreasing Blood Loss Prior to Abdominal Myomectomy: A Randomized Double-blinded Clinical Trial
Brief Title: Sublingual Misoprostol in Decreasing Blood Loss Prior to Myomectomy
Acronym: SL-MISO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: misop 2
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Blood Loss in Myomectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Placebo Comparator): 400 mg placebo
  Interventions: Drug: placebo 400 sublingual
- Group B (Active Comparator): 400 microgram misoprostol
  Interventions: Drug: Misoprostol 400 sublingual

INTERVENTIONS:
Drug: Misoprostol 400 sublingual — patients will take 2 tablets of sublingual misoprostol 400 microgram 3 hours and 1 hour before the surgery
  Arms: Group B
Drug: placebo 400 sublingual — patients will take 2 tablets of sublingual placebo 400 microgram 1 hour before the surgery
  Arms: Group A

SUMMARY:
The aim of the study is to compare the effectiveness of sublingual administered prostaglandin E1 synthetic analogue (misoprostol) 400 microgram versus placebo before myomectomy to decrease blood loss during and after the operation.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for abdominal myomectomy with documented uterine fibroids on pelvic imaging
* Age ≥ 18 years and ≤ 50 years
* Pre-operative hemoglobin >8 g/dl
* Ability to understand and the willingness to sign a written informed consent.
* Admissible medical/surgical history
* Five or less symptomatic uterine myomas
* All myomas are subserous or intramural.
* Uterine size less than 24 weeks pregnancy

Exclusion Criteria:

* Patients who have had a prior abdominal myomectomy
* Post-menopausal women
* Patients with known bleeding/clotting disorders
* Patients with a history of gynecologic malignancy
* Hypertension.
* Cardiac and Pulmonary diseases.
* Obesity (body mass index > 30 kg/m2).
* History of allergic reactions attributed to misoprostol
* Cases that will require intraoperative conversion of myomectomy to hysterectomy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Mean amount of intraoperative blood loss | intraoperative

SECONDARY OUTCOMES:
Change of hemoglobin after surgery | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No